CLINICAL TRIAL: NCT00401583
Title: A Multi-center, Open-Label, Multiple-probe Drug Interaction Study to Determine the Effects of GW786034 on the Metabolism of Cytochrome P450 Probe Drugs in Patients With Solid Tumors
Brief Title: A Study To Test The Effect Of GW786034 (Pazopanib) On P450 Enzymes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG10007
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: GW786034 (pazopanib) cytochrome P450 interaction
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib receivers (Experimental): During Days 1 and 2 subjects will be dosed with only probe drugs, and with no drugs on Days 3-5. During Days 6 to the end of the study, subjects will receive 800 mg daily pazopanib, and on Days 23-24 subjects will receive probe drugs in addition to pazopanib
  Interventions: Drug: GW786034 (pazopanib); Drug: Probe drugs

INTERVENTIONS:
Drug: GW786034 (pazopanib) — Pazopanib will be given as monohydrochloride, 100 and 500 mg tablets.
Drug: Probe drugs — probe drugs will be oral midazolam (3 mg), warfarin (10 mg), omeprazole (40 mg), caffeine (200 mg), and dextromethorphan (30 mg).

SUMMARY:
This is a Phase I study to determine the effect of GW786034 (pazopanib) on P450 enzymes. This study will help determine which types of drugs may interact with GW786034.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumors.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone marrow, renal, lung, and liver function.
* A female subject must not be pregnant and will agree not to become pregnant during the trial

Exclusion criteria:

* Any major surgery, chemotherapy, hormone therapy, investigational drugs, or radiotherapy within the last 28 days.
* Poorly controlled hypertension.
* Corrected QT (QTc) prolongation defined as a QTc interval greater than or equal to 480 msec and a prior history of cardiovascular disease, arrhythmias, or significant ECG abnormalities.
* Arterial or venous thrombi (including cerebrovascular accident), myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within the last 3 months.
* Current use of therapeutic anticoagulation (low molecular weight heparin, oral anticoagulant agents).

Amiodarone must not have been taken for at least 6 months prior to the administration of the first dose of study drug.

* History of brain metastases.
* Has narrow-angle glaucoma which is a contraindication to midazolam use.
* History of nicotine-containing product (including cigarettes, cigars, nicotine patches) use within the past 6 months.
* A history of bleeding problems.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-07-28 (Actual); Primary Completion 2008-02-20 (Actual); Study Completion 2008-02-20 (Actual)

PRIMARY OUTCOMES:
To investigate the potential of GW786034 to inhibit or induce various CYP450 enzymes. | throughout the study

SECONDARY OUTCOMES:
Safety of co-administration of 800 mg daily GW786034 and CYP450 probe drugs. To describe GW786034 steady-state pharmacokinetics on this once daily dosing regimen. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Lebanon, New Hampshire, United States
- GSK Investigational Site, Singapore, Singapore

REFERENCES:
- [Background] Goh BC, Reddy NJ, Dandamudi UB, Laubscher KH, Peckham T, Hodge JP, Suttle AB, Arumugham T, Xu Y, Xu CF, Lager J, Dar MM, Lewis LD. An evaluation of the drug interaction potential of pazopanib, an oral vascular endothelial growth factor receptor tyrosine kinase inhibitor, using a modified Cooperstown 5+1 cocktail in patients with advanced solid tumors. Clin Pharmacol Ther. 2010 Nov;88(5):652-9. doi: 10.1038/clpt.2010.158. Epub 2010 Sep 29. PMID 20881954
- See also: Results for study VEG10007 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/VEG10007?search=study&search_terms=VEG10007#rs